CLINICAL TRIAL: NCT02273336
Title: Genomics of Young Lung Cancer Study
Brief Title: Comprehensive Genomic Analysis in Tissue and Blood Samples From Young Patients With Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: Foundation Medicine (Industry); Addario Lung Cancer Medical Institute (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ALCMI-003; NCI-2014-02098 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2L-14-1; ALCMI-003 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-10-21; First posted 2014-10-23 (Estimated); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Non-small Cell Lung Cancer; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (comprehensive genomic analysis): Tissue and blood samples are analyzed via next generation sequencing and whole exome sequencing.
  Interventions: Other: cytology specimen collection procedure; Other: laboratory biomarker analysis

INTERVENTIONS:
Other: cytology specimen collection procedure — Undergo tissue and blood sample collection
  Other Names: cytologic sampling
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This research trial studies genomic analysis in tissue and blood samples from young patients with lung cancer. Identifying specific gene mutations (changes in deoxyribonucleic acid [DNA]) may help doctors tailor treatment to target the specific mutations and help plan effective treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform comprehensive genomic analysis of young lung cancer patients' samples to facilitate delivery of targeted therapies and clinical trial enrollment.

II. To characterize the impact of young age at lung cancer diagnosis on the genomic landscape of primary lung cancer.

III. To establish a prospective registry of young lung cancer patients for both tumor and germline next generation sequencing.

OUTLINE:

Tissue and blood samples are analyzed via next generation sequencing and whole exome sequencing.

After completion of study, patients are followed up every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* COHORT 1: LUNG CANCER PATIENTS
* Pathologically confirmed bronchogenic lung carcinoma (small cell lung cancer [SCLC] or non-small cell lung cancer [NSCLC] of any stage) at any treatment time point
* For individuals diagnosed with advanced disease (stage IV or recurrent) enrollment must occur within 2 years of diagnosis
* For appropriate patients (stage IV non-squamous NSCLC) epidermal growth factor receptor (EGFR ) and anaplastic lymphoma kinase (ALK) genotyping performed by a Clinical Laboratory Improvement Amendments (CLIA) certified laboratory is recommended prior to participation
* Provision of written informed consent
* Willingness to undergo a single blood draw
* Individuals who are under 18 are eligible for study if they meet the defined criteria for cohort 1; in addition, consent for participation must be given by a legal guardian or parent

  * NOTE: to be eligible for genomics, availability of 10 unstained slides (plus hematoxylin and eosin [H&E] slide) or an adequate formalin-fixed paraffin-embedded (FFPE) tumor block from clinically indicated interventional procedures is required
* COHORT 2: DECEASED INDIVIDUALS
* Deceased individuals diagnosed with lung cancer at any age less than 40 may be studied on a case by case basis depending upon Institutional Review Board (IRB) approval at a participating institution; inclusion will require availability of adequate archived FFPE tissue and release of tissue and records by next of kin, if available

Exclusion Criteria:

* Compromise of patient diagnosis or staging if tissue is used for research

Max Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects will be recruited at Dana Farber Institute and USC Norris Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-07-22 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Prevalence of targetable mutations, defined as any alteration in a drive oncogene for which Food and Drug Administration-approved therapy exists, for which an off-label therapy exists, or for which a clinical trial exists | Baseline
  Will compare this population with the historical experience of the Lung Cancer Mutation Consortium. For this specific comparison, the prevalence of mutations in EGFR, ALK, v-raf murine sarcoma viral oncogene homolog B1 (BRAF), human epidermal growth factor receptor 2 (HER2), v-ros avian UR2 sarcoma virus oncogene homolog 1 (ROS1), and met proto-oncogene (MET) will be calculated.
Proportion of young lung cancer patients that enroll onto clinical trials | Baseline
Proportion of patients that received targeted therapies based on their clinical genotyping results | Baseline
Acquired deactivating mutations | Baseline
  All data summaries based on next generation sequencing of tumor and blood deoxyribonucleic acid/ribonucleic acid will be descriptive, with the goal of discovering novel tumor suppressor genes that may be deactivated leading to the development of NSCLC in individuals less than 40 years.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gitlitz, MD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Dana-Farber Cancer Institute, Boston, Massachusetts